CLINICAL TRIAL: NCT02243709
Title: A Pilot Study on the Safety and Efficacy of Mifepristone for the Prevention of Relapses of Alcohol Drinking
Brief Title: Mifepristone for the Prevention of Relapses of Alcohol Drinking
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Carolina L Haass-Koffler, Research Fellow, Brown University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1404001031
Record Dates: First submitted 2014-09-12; First posted 2014-09-18 (Estimated); Results first posted 2023-06-01 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorders (AUD)
Keywords: Stress, alcohol craving, alcohol use disorders
MeSH Terms: conditions — Alcoholism | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mifepristone (Active Comparator): mifepristone 600-mg/day for a week, in a stress-induced condition triggered by a single dose of 32.4-mg of yohimbine
  Interventions: Drug: Mifepristone 600-mg/day or placebo for a week
- Sugar pill (Placebo Comparator): matching placebo/day for a week, in a stress-induced condition triggered by a single dose of 32.4-mg of yohimbine
  Interventions: Drug: Mifepristone 600-mg/day or placebo for a week

INTERVENTIONS:
Drug: Mifepristone 600-mg/day or placebo for a week — 600-mg of mifepristone for a week, compared to placebo for a week, in a stress-induced condition triggered by a single dose of 32.4 mg of yohimbine

SUMMARY:
The goal of this study is to determine if, under stress, alcohol drinking is reduced using mifepristone

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 21 to 65 years of age
* Females must be postmenopausal for at least one year or surgically sterile (proven by medical record)
* Meet criteria for Alcohol Use Disorders (AUD) DSM-5 diagnosis
* Meet drinking criteria (≥3 drinks/day for men; ≥2 drinks /day for women)
* Must be in good health as confirmed by medical history, physical examination, ECG, lab tests
* Participants must be willing to take oral medication and adhere to the study procedures
* Breath alcohol (BrAC) = 0.00 at each visit
* Be able to understand informed consent and questionnaire in English at an 8th grade level

Exclusion Criteria:

* Individuals expressing interest in treatment for alcoholism
* Premenopausal women
* Participants who have significant alcohol withdrawal symptoms, defined as a CIWA-Ar score ≥7
* A repeated positive urine drug screen at baseline for any illegal substance except marijuana.
* Individuals diagnosed with a current "severe" Substance Use Disorder (SUD) diagnosis, other than alcohol or nicotine
* Meet DSM-5 criteria for a diagnosis of schizophrenia, bipolar disorder, or other psychoses
* An active illness within the past six months of the screening visit that meets the DSM-5 criteria for a diagnosis of Major Depressive Disorder (MDD) or Anxiety Disorder, or history of attempted suicide
* Clinically significant medical abnormalities: unstable hypertension, clinically significant abnormal ECG, bilirubin >150% of the upper normal limit, ALT/AST >300% the UNL, creatinine clearance ≤60 dl/min
* Current use of psychotropic medications that may have an effect on alcohol consumption
* Current use of any medication involved in the metabolism of alcohol such as aldehyde dehydrogenase (ALDH), alcohol dehydrogenase (ADH) and CYP2E1: Cefamandole, Cefotetan, Sulfamethoxazole, Nitroglycerin, Chlorpropamide, Glyburide.
* Current use of any medication (CYP3A4 inhibitor and substrate) that may interact with mifepristone: cyclosporine, fentanyl, heparin, escitalopram, lovastatin, simvastatin, warfarin
* Current use of any medication (CYP2D6 inhibitor and substrate) that may interact with yohimbine: amitriptyline, doxepin, nortriptyline, venlafaxine
* Medical contraindications for use of mifepristone or yohimbine
* A history of adverse reaction or hypersensitivity to mifepristone or yohimbine
* History of suicide
* History of seizure disorders
* Hypokalemia (low potassium level)<3.5mEq/L
* Participated in any behavioral and/or pharmacological study within minimum the past 30 days
* Neuroendocrine disorders
* Taking corticosteroids
* Bleeding disorders
* Pre-existing QT prolongation on ECG
* History of porphyria (Mifepristone progesterone receptor antagonist is an inducer of CYP-450 and therefore may have the ability to precipitate or exacerbate attacks of acute porphyria)
* Not willing to engage in protected sex (condom). This risk includes both women and men. Mifepristone long half-life (t1/2 = 18 hrs) and its three main metabolites retain considerable affinity toward human progesterone and glucocorticoid receptors, with serum level similar to the parent mifepristone and there are no studies on the presence of mifepristone or metabolites in semen

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina L Haass-Koffler, PharmD, Principal Investigator — Brown University
Locations (1):
- Center for Alcohol and Addiction Studies, Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Result] Simms JA, Haass-Koffler CL, Bito-Onon J, Li R, Bartlett SE. Mifepristone in the central nucleus of the amygdala reduces yohimbine stress-induced reinstatement of ethanol-seeking. Neuropsychopharmacology. 2012 Mar;37(4):906-18. doi: 10.1038/npp.2011.268. Epub 2011 Nov 2. PMID 22048462
- [Result] Haass-Koffler CL, Magill M, Cannella N, Brown JC, Aoun EG, Cioe PA, Sinha R, Swift RM, Ciccocioppo R, Leggio L. Mifepristone as a pharmacological intervention for stress-induced alcohol craving: A human laboratory study. Addict Biol. 2023 Jul;28(7):e13288. doi: 10.1111/adb.13288. PMID 37369125
- [Derived] Haass-Koffler CL, Magill M, Cannella N, Brown JC, Aoun EG, Cioe PA, Sinha R, Swift RM, Ciccocioppo R, Leggio L. Mifepristone as a pharmacological intervention for stress-Induced alcohol craving: a translational crossover randomized trial. medRxiv [Preprint]. 2023 Jan 4:2023.01.02.23284122. doi: 10.1101/2023.01.02.23284122. PMID 36711869

RESULTS

PARTICIPANT FLOW:
Groups:
- Mifepristone, Then Placebo: Participants receive mifepristone 600-mg/day for one week. Participants then go through a 3 week wash out period where no medications are dispensed. Participants then receive a matched placebo (matching Mifepristone) for one week.
- Placebo, Then Mifepristone: Participants receive a placebo pill for one week. Participants then go through a 3 week wash out period where no medications are dispensed. Participants then receive a matched Mifepristone (600 mg/day) dose for one week.
Period: Phase 1
Arm/Group | Mifepristone, Then Placebo | Placebo, Then Mifepristone
Started | 12 | 20
Completed | 11 | 17
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Phase 2: Crossover to Opposite Condition
Arm/Group | Mifepristone, Then Placebo | Placebo, Then Mifepristone
Started | 11 | 17
Completed | 11 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Sample: All participants receive either Mifepristone (600 mg) or matched placebo that is randomized within a cross-over, double blind clinical trial.
Arm/Group | Overall Sample
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 9
  WHITE | 22
  Multiracial | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32
Alcohol craving [Mean (Standard Deviation); unit: units on a scale] — Alcohol craving will be assessed by the Alcohol Craving Questionnaire Short Form - Revised (ACQ-SF-R). The ACQ-SF-R is a 12-item self-report scale that contains items from the 47-item Alcohol Craving Questionnaire (ACQ-Now). ACQ-SF-R also produces scores for compulsivity, expectancy, purposefulness, and emotionality. In this study, at baseline/the first study visit, the 12-item total ACQ will be summed for each participant and then the total score will be averaged for a mean score. The ACQ has a total score range between 0-84. A lower score indicates less subjective alcohol craving.
  units on a scale | 40.9 (14.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events in the Mifepristone Versus Placebo Group as a Measure of Safety and Tolerability
Description: Safety and tolerability was assessed by the number of participants who experienced adverse events (AEs) while taking the medication, in the mifepristone group verses the placebo group during Visit 2 through and until Visit 5. AEs were assessed at each visit and special attention was paid to any AEs experienced after administration of the oral administration of mifepristone or placebo- Visit 2 to Visit 3 (7 days total) and Visit 4 through Visit 5 (7 days total), and when it was administered with alcohol during the laboratory paradigms at visits 3 and 4.
Time Frame: 5 weeks (one week of drug administration, 3 weeks of washout, followed by one week of drug administration)
Measure: Count of Participants; unit: Participants
Groups:
- Mifepristone: mifepristone 600-mg/day for a week, after a single dose of 32.4-mg of yohimbine
- Placebo: matching placebo/day for a week, after a single dose of 32.4-mg of yohimbine
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 27 | 31
Participants | 0 | 3
Statistical Analysis 1: Comparison: Mifepristone vs Placebo; Test type: Other; p > .05, Chi-squared

2. Secondary Outcome: Alcohol Craving Score on the Alcohol Craving Questionnaire in the Mifepristone Versus Placebo Group
Description: Alcohol craving will be assessed by the Alcohol Craving Questionnaire Short Form - Revised (ACQ-SF-R). The ACQ-SF-R is a 12-item self-report scale that contains items from the 47-item Alcohol Craving Questionnaire (ACQ-Now). ACQ-SF-R also produces scores for compulsivity, expectancy, purposefulness, and emotionality. To assess this outcome, at the alcohol cue reactivity procedures/visits 3 and 5 during alcohol trial 1, the 12-item total ACQ will be summed for each participant and then the total score will be averaged for a mean score. The average ACQ score in the presence of alcohol cues will be compared when participants are taking mifepristone compared to placebo. The ACQ has a total score range between 0-84. A lower score indicates less subjective alcohol craving.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mifepristone: Mifepristone 600-mg/day for one week.
- Placebo: Administration of matched placebo for one week.
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 27 | 31
score on a scale | 42.92 (17.85) | 50.13 (19.3)

3. Secondary Outcome: Drinking Consumption in the Mifepristone Verses Placebo Group
Description: Number of standard drinks desired to be consumed by participants during mifepristone administration compared to placebo administration during the open bar (free choice procedure) in the alcohol cue reactivity at visits 3 and 5.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: drinks
Groups:
- Mifepristone: Administration of mifepristone 600-mg/day for one week.
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 27 | 31
drinks | 0.8 (0.3) | 0.5 (0.2)

ADVERSE EVENTS:
Time Frame: AEs were monitored for 5 weeks (one week of medication administration, followed by a three week wash out period, then followed by another week of medication administration). Medication administration is randomized between subjects within a cross over design.
Description: Participant were screened initially with a full physical assessment
Arm/Group | Mifepristone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/31
Other Adverse Events (participants affected / at risk) | 0/27 | 3/31
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=27) | Placebo (N=31)
emesis (Gastrointestinal disorders) | 0 (0) | 2 (2)
hypertension (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-12-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT02243709/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT02243709/SAP_001.pdf